CLINICAL TRIAL: NCT02059434
Title: A 2-Part, Randomised, Placebo-Controlled, Safety, Tolerability, Pharmacokinetic And Pharmacodynamic Study Of LAS190792 Delivered By Inhalation In Asthmatic And Chronic Obstructive Pulmonary Disease (COPD) Subjects
Brief Title: Two-part Pharmacokinetic and Pharmacodynamic Study of LAS190792 in Patients With Asthma and COPD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: M-190792-01; 2013-001758-93 (EudraCT Number)
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Tiotropium Bromide; indacaterol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (12):
- LAS190792 Dose 1 (Part 1) (Experimental): Single dose, oral inhalation by Genuair® single-dose dry powder inhaler (DPI)
  Interventions: Drug: LAS190792 Dose 1
- LAS190792 Dose 2 (Part 1) (Experimental): Single dose, oral inhalation by Genuair® single-dose dry powder inhaler (DPI)
  Interventions: Drug: LAS190792 Dose 2
- LAS190792 Dose 3 (Part 1) (Experimental): Single dose, oral inhalation by Genuair® single-dose dry powder inhaler (DPI)
  Interventions: Drug: LAS190792 Dose 3
- LAS190792 Dose 4 (Part 1) (Experimental): Single dose, oral inhalation by Genuair® single-dose dry powder inhaler (DPI)
  Interventions: Drug: LAS190792 Dose 4
- LAS190792 Dose 5 (Part 1) (Experimental): Single dose, oral inhalation by Genuair® single-dose dry powder inhaler (DPI)
  Interventions: Drug: LAS190792 Dose 5
- LAS190792 Dose 6 (Part 1) (Experimental): Single dose, oral inhalation by Genuair® single-dose dry powder inhaler (DPI)
  Interventions: Drug: LAS190792 Dose 6
- Placebo (Part 1) (Placebo Comparator): Single dose, oral inhalation by Genuair® single-dose dry powder inhaler (DPI)
  Interventions: Drug: Placebo
- LAS190792 Dose 1 (Part 2) (Experimental): Single dose, oral inhalation by Genuair® single-dose dry powder inhaler (DPI)
  Interventions: Drug: LAS190792 Dose 1 (Part 2)
- LAS190792 Dose 2 (Part 2) (Experimental): Single dose, oral inhalation by Genuair® single-dose dry powder inhaler (DPI)
  Interventions: Drug: LAS190792 Dose 2 (Part 2)
- Tiotropium 18 μg (Active Comparator): Single dose, oral inhalation by HandiHaler® single-dose DPI
  Interventions: Drug: Tiotropium 18 μg
- Indacaterol 150 μg (Active Comparator): Single dose, oral inhalation by Breezhaler® single-dose DPI
  Interventions: Drug: Indacaterol 150 μg
- Placebo (Part 2) (Placebo Comparator): Single dose, oral inhalation by Genuair® single-dose dry powder inhaler (DPI)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LAS190792 Dose 1
  Arms: LAS190792 Dose 1 (Part 1)
Drug: LAS190792 Dose 2
  Arms: LAS190792 Dose 2 (Part 1)
Drug: LAS190792 Dose 3
  Arms: LAS190792 Dose 3 (Part 1)
Drug: LAS190792 Dose 4
  Arms: LAS190792 Dose 4 (Part 1)
Drug: LAS190792 Dose 5
  Arms: LAS190792 Dose 5 (Part 1)
Drug: LAS190792 Dose 6
  Arms: LAS190792 Dose 6 (Part 1)
Drug: LAS190792 Dose 1 (Part 2)
  Arms: LAS190792 Dose 1 (Part 2)
Drug: LAS190792 Dose 2 (Part 2)
  Arms: LAS190792 Dose 2 (Part 2)
Drug: Tiotropium 18 μg
  Other Names: Spiriva
  Arms: Tiotropium 18 μg
Drug: Indacaterol 150 μg
  Other Names: Onbrez
  Arms: Indacaterol 150 μg
Drug: Placebo
  Arms: Placebo (Part 1); Placebo (Part 2)

SUMMARY:
The purpose of this study is to assess the safety and tolerability of single doses of LAS190792 administered by inhalation to patients with mild persistent asthma and moderate to severe chronic obstructive pulmonary disease (COPD) and also to assess the ability of LAS190792 to produce bronchodilation (opening of the airways).

DETAILED DESCRIPTION:
This study is an integrated Phase I protocol divided into 2 parts.

Part one: a single ascending dose study (6 LAS190792 dose levels) in 16 male subjects with mild asthma. LAS190792 will be administered (by the Genuair® inhaler) under supervision at the study centre, according to the randomisation scheme. One dose level will be administered per week with 2 to 3 weeks between each dose level for the safety and pharmacokinetic data review.

Part two: A 5-way , crossover, single dose study (of LAS190792 [two doses], indacaterol, tiotropium and placebo) in 40 male and non-childbearing potential women subjects with moderate to severe COPD. Each treatment period will be separated by a washout period of at least 7 to 14 days. The aim is to ensure at least 30 subjects complete Part 2 of the study. The primary comparison for bronchodilation will be between LAS190792 doses and placebo. Other treatment comparisons (indacaterol or tiotropium vs placebo and LAS190792 vs indacaterol or tiotropium) will be considered additional.

ELIGIBILITY:
Inclusion Criteria (PART 1):

* Adult male subjects aged 18 to 70 years
* Body mass index (BMI) 18.5 to 30 kg/m2 at screening
* Clinical diagnosis of mild persistent asthma (according to GINA guidelines) for at least 6 months prior to screening
* Ability to change current asthma therapy, to discontinue previous prescribed medications after signature of informed consent as per required washout periods
* Screening FEV1 value of ≥70% of the predicted normal value after a washout of at least 5 h for short-acting beta2-agonists and 72 h for long-acting beta2-agonists
* FEV1 reversibility of ≥12% and an absolute increase of at least 200 mL over the baseline value within 30 min after inhalation of 400 µg of salbutamol
* Subjects using intermittent salbutamol and / or subjects on a stable dose or regimen of low dose ICS (as defined by the GINA guidelines) at least 4 weeks prior to screening
* Predose FEV1 value of first treatment period within the range of ±20% of the FEV1 measured at screening prior to salbutamol inhalation
* Subjects who are otherwise healthy as determined by medical history, physical examination, 12-lead ECG findings
* Normal blood pressure (defined as SBP between 100 and 140 mmHg, and DBP between 50 and 90 mmHg) at screening, measured after resting in supine position for 5 minutes.
* Subjects whose clinical laboratory test results are not clinically relevant and are acceptable to the Investigator
* Subjects who are negative for hepatitis B surface antigen (HBsAg), hepatitis B core (HBc) antibody (IgM), hepatitis C antibody and human immunodeficiency virus (HIV) I and II antibodies at screening
* Subjects who are able and willing to provide written informed consent
* Subjects able to perform repeatable pulmonary function testing for FEV1 according to the American Thoracic Society (ATS) / European Respiratory Society (ERS) 2005 criteria at screening

Inclusion Criteria (PART 2):

* Adult male and non-childbearing potential women subjects aged ≥40 years with a clinical diagnosis of stable moderate to severe COPD according to GOLD guidelines at screening
* Females must be of non-childbearing potential, confirmed at screening
* Post-salbutamol FEV1 <80% and ≥30% of the predicted normal value and post-salbutamol FEV1 / forced vital capacity (FVC) <70%
* Ability to change current COPD therapy, to discontinue previous prescribed medications after signature of informed consent
* No evidence of clinically significant respiratory and / or cardiovascular conditions or laboratory abnormalities
* No other relevant pulmonary disease or history of thoracic surgery
* No contraindication to the use of anticholinergic drugs such as known symptomatic prostatic hypertrophy, bladder neck obstruction, narrow-angle glaucoma, or beta2-agonists usage
* Subjects who are negative for HBsAg, HBc IgM, hepatitis C antibody and HIV I and II antibodies at screening
* Subjects who are able and willing to provide written informed consent
* Subjects able to perform repeatable pulmonary function testing for FEV1 according to the ATS / ERS 2005 criteria at screening

Exclusion Criteria (PART 1 and 2):

* Subjects who do not conform to the above inclusion criteria
* Current smokers, subjects with a smoking history during the last 12 months or subjects with a smoking history of more than 10 pack-years
* Other relevant pulmonary disease or history of thoracic surgery
* Subjects with a BMI ≥40 kg/m2 (only applicable for Part 2)
* Subjects with any clinically relevant history or presence of abnormality from the medical history and/or physical examination (only applicable for Part 1)
* Current evidence or recent history of any clinically significant and unstable disease (other than COPD) or abnormality that could put the subject at risk or could confound the results of the study (only applicable for Part 2)
* Subjects with a surgical history clinically relevant for the purpose of the study
* History of malignancy of any organ system, treated or untreated within the past 5 years, with the exception of localised basal cell carcinoma of the skin
* Subjects with serious adverse reaction or serious hypersensitivity to Spiriva (for Part 2 only), indacaterol (for Part 2 only), or the formulation excipients (eg, lactose) or other drugs in the same pharmacologic class (for Part 1 and Part 2)
* Current diagnosis of COPD (for Part 1 only) or history of / or current diagnosis for asthma (for Part 2 only)
* Recent history of asthma / COPD exacerbation requiring hospitalisation or need for increased maintenance treatments for asthma / COPD within 6 weeks prior to screening or randomisation
* Use of daily oxygen therapy >10 h per day (for Part 2 only)
* Use of systemic steroids for respiratory reasons within 3 months prior to screening
* Lower respiratory tract infection within 6 weeks prior to screening or randomisation
* Upper respiratory tract infection requiring antibiotics within 4 weeks prior to screening or randomisation
* Current history of tuberculosis, bronchiectasis or other non-specific pulmonary disease
* QTcF interval >430 ms at screening or prior to randomisation, or history of long QT syndrome (for Part 1 only)
* QTcF interval, >450 ms for males and >470 ms for females at screening or prior to randomisation, or history of long QT syndrome (for Part 2 only)
* Subjects with a history of excessive use or abuse of alcohol or with a history of drug abuse within the past 2 years
* Subjects who are positive for drugs of abuse and alcohol tests at screening and prior to randomisation
* Donation or loss >400 ml of blood and plasma within the previous 3 months prior to screening
* Subjects consuming more than 14 (female subjects) or 21 (male subjects) units of alcohol a week
* Subjects with a significant infection or known inflammatory process at screening or prior to randomisation
* Subjects with acute gastrointestinal symptoms at the time of screening or prior to randomisation
* Subjects with an acute infection such as influenza at the time of screening or prior to randomisation
* Male subjects who do not agree to follow instructions to avoid pregnancies
* Subjects who are not able to adhere to the restrictions on prior and concomitant medications
* Subjects who intend to use any concomitant medication not permitted by the protocol or who have not undergone the required washout period for a particular prohibited medication
* Subjects who have used any investigational drug within 3 months prior to screening or within the equivalent time of 6 half-lives of receiving the last administration, whichever is longer
* Subjects who have received the last dose of investigational product more than 3 months ago but who are on an extended follow-up
* Subjects who are vegans or who have medical dietary restrictions
* Subjects unable to communicate reliably with the Investigator
* Subjects who are unlikely to co-operate with the requirements of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2014-10-06 (Actual); Study Completion 2014-10-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Quintiles Drug Research Unit at Guy's Hospital, London
  - Medicines Evaluation Unit Ltd (MEU), Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 centres in the UK. In part 1 of the study, the first patient was screened in September 2013 and the last patient visit was in February 2014. In part 2 of the study, the first patient was screened in March 2014 and the last patient visit was in October 2014.
Pre-assignment Details: This was a 2-part study.
  Part 1: incomplete crossover, single ascending dose study of 2 cohorts randomised to fixed sequences of LAS190792 or placebo in 3 treatment periods.
  Part 2: 5-way complete crossover, single dose study of LAS190792 (100/400 μg), placebo, or active controls (indacaterol 150 μg, tiotropium 18 μg) in 5 treatment periods.
Groups:
- Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg: All individuals in Part 1 - Cohort 1 who were randomised to treatment sequence LAS190792 5 μg, 50 μg, 200 μg in 3 treatment periods separated by washout periods of 28-42 days.
- Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg: All individuals in Part 1 - Cohort 1 who were randomised to treatment sequence Placebo, then LAS190792 50 μg, 200 μg in 3 treatment periods separated by washout periods of 28-42 days.
- Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg: All individuals in Part 1 - Cohort 1 who were randomised to treatment sequence LAS190792 5 μg, Placebo, LAS190792 200 μg in 3 treatment periods separated by washout periods of 28-42 days.
- Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo: All individuals in Part 1 - Cohort 1 who were randomised to treatment sequence LAS190792 5 μg, 50 μg, then Placebo in 3 treatment periods separated by washout periods of 28-42 days.
- Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg: All individuals in Part 1 - Cohort 2 who were randomised to treatment sequence LAS190792 20 μg, 100 μg, 400 μg in 3 treatment periods separated by washout periods of 28-42 days.
- Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg: All individuals in Part 1 - Cohort 2 who were randomised to treatment sequence Placebo, then LAS190792 100 μg, 400 μg in 3 treatment periods separated by washout periods of 28-42 days.
- Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg: All individuals in Part 1 - Cohort 2 who were randomised to treatment sequence LAS190792 20 μg, Placebo, LAS190792 400 μg in 3 treatment periods separated by washout periods of 28-42 days.
- Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo: All individuals in Part 1 - Cohort 2 who were randomised to treatment sequence LAS190792 20 μg, 100 μg, then Placebo in 3 treatment periods separated by washout periods of 28-42 days.
- Overall Population - Part 2: All individuals involved in Part 2 (single-dose study of two doses of LAS190792 [100 and 400 μg], indacaterol, tiotropium or placebo, in 5 treatment periods separated by washout periods of 7-14 days).
Period: Period 1 (After Screening/run-in Period)
Arm/Group | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg | Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg | Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo | Overall Population - Part 2
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 0 (Part 2 followed Part 1, and comprised 5 treatment periods)
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 0 (Part 2 followed Part 1, and comprised 5 treatment periods)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Between Periods 1 and 2
Arm/Group | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg | Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg | Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo | Overall Population - Part 2
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 0 (Part 2 followed Part 1, and comprised 5 treatment periods)
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 (Part 2 followed Part 1, and comprised 5 treatment periods)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg | Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg | Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo | Overall Population - Part 2
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 (Part 2 followed Part 1, and comprised 5 treatment periods)
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 (Part 2 followed Part 1, and comprised 5 treatment periods)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Between Periods 2 and 3
Arm/Group | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg | Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg | Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo | Overall Population - Part 2
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 (Part 2 followed Part 1, and comprised 5 treatment periods)
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 (Part 2 followed Part 1, and comprised 5 treatment periods)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg | Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg | Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo | Overall Population - Part 2
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 (Part 2 followed Part 1, and comprised 5 treatment periods)
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 (Part 2 followed Part 1, and comprised 5 treatment periods)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4 (After Screening/run-in Period)
Arm/Group | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg | Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg | Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo | Overall Population - Part 2
Started | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 38
Completed | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 38
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Between Periods 4 and 5
Arm/Group | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg | Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg | Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo | Overall Population - Part 2
Started | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 38
Completed | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 37
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 5
Arm/Group | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg | Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg | Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo | Overall Population - Part 2
Started | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 37
Completed | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 37
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Between Periods 5 and 6
Arm/Group | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg | Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg | Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo | Overall Population - Part 2
Started | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 37
Completed | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 37
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 6
Arm/Group | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg | Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg | Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo | Overall Population - Part 2
Started | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 37
Completed | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 37
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Between Periods 6 and 7
Arm/Group | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg | Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg | Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo | Overall Population - Part 2
Started | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 37
Completed | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 36
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 7
Arm/Group | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg | Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg | Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo | Overall Population - Part 2
Started | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 36
Completed | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 36
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Between Periods 7 and 8
Arm/Group | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg | Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg | Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo | Overall Population - Part 2
Started | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 36
Completed | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 34
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 8
Arm/Group | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg | Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg | Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo | Overall Population - Part 2
Started | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 34
Completed | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 0 (Part 1 comprised 3 treatment periods only) | 34
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of participants randomised in Part 1 - Cohorts 1 and 2 treatment sequences (incomplete crossover design) and overall in Part 2 (due to 5-way crossover design), respectively.
  Parts 1 and 2 were independent: there was no intention to compare the results of the 2 parts of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, 200 μg | Part 1 - Cohort 1 Placebo, Then LAS190792 50 μg, 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, Placebo, LAS190792 200 μg | Part 1 - Cohort 1 LAS190792 5 μg, 50 μg, Then Placebo | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, 400 μg | Part 1 - Cohort 2 Placebo, Then LAS190792 100 μg, 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, Placebo, LAS190792 400 μg | Part 1 - Cohort 2 LAS190792 20 μg, 100 μg, Then Placebo | Overall Population - Part 2 | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 38 | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Baseline characteristics for participants randomised in Part 1 - Cohorts 1 and 2 treatment sequences (incomplete crossover design) and overall in Part 2 (due to 5-way crossover design), respectively.
  Years
    Part 1: number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 0 | 17
    Part 1 | 35 (8.5) | 34.5 (20.5) | 35 (4.2) | 37 (19.8) | 32.5 (6.4) | 41.5 (29.0) | 28 (1.4) | 34.3 (12.7) |  | 34.7 (12.0)
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 38 | 38
    Part 2 |  |  |  |  |  |  |  |  | 60.4 (5.9) | 60.4 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics for participants randomised in Part 1 - Cohorts 1 and 2 treatment sequences (incomplete crossover design) and overall in Part 2 (due to 5-way crossover design), respectively.
  Participants
    Part 1: number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 0 | 17
    Part 1: Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part 1: Male | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 0 | 17
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 38 | 38
    Part 2: Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18
    Part 2: Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 20

OUTCOME MEASURES:

1. Primary Outcome: Subjects With ≥1 Treatment-emergent Adverse Event
Description: Adverse events (AEs) are any unfavorable and unintended medical occurrence during the subject's participation in the study (including deterioration of a pre-existing medical condition, an abnormal value in a laboratory assessment, an ECG abnormality, a 12-lead 24-hour ECG-Holter abnormality, a blood pressure abnormal value, paradoxal bronchospasm or an abnormal finding in the physical examination) and will be coded using the current Medical Dictionary for Regulatory Activities (MedDRA).
Time Frame: 30 Days
Population: Safety Population: defined as all randomized subjects who received at least one dose of the investigational product
Measure: Number; unit: Participants
Groups:
- LAS190792 5 µg (Part 1); LAS190792 20 µg (Part 1); LAS190792 50 µg (Part 1); LAS190792 100 µg (Part 1); LAS190792 200 µg (Part 1); LAS190792 400 µg (Part 1); Placebo (Part 1); LAS190792 100 µg (Part 2); LAS190792 400 µg (Part 2); Placebo (Part 2): Single dose, oral inhalation by Genuair® single-dose dry powder inhaler (DPI)
- Tiotropium 18 μg: Single dose, oral inhalation by HandiHaler® single-dose dry powder inhaler (DPI)
- Indacaterol 150 μg: Single dose, oral inhalation by Breezhaler® single-dose dry powder inhaler (DPI)
Arm/Group | LAS190792 5 µg (Part 1) | LAS190792 20 µg (Part 1) | LAS190792 50 µg (Part 1) | LAS190792 100 µg (Part 1) | LAS190792 200 µg (Part 1) | LAS190792 400 µg (Part 1) | Placebo (Part 1) | LAS190792 100 µg (Part 2) | LAS190792 400 µg (Part 2) | Tiotropium 18 μg | Indacaterol 150 μg | Placebo (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 36 | 35 | 37 | 37 | 37
Participants | 2 | 3 | 2 | 2 | 2 | 4 | 3 | 12 | 12 | 14 | 21 | 15

2. Primary Outcome: Change From Baseline in Trough FEV1 (Forced Expiratory Volume in 1 Second)
Description: Trough is defined as the mean of the FEV1 values obtained at 23 hours and at 24 hours after morning investigational product administration.
Time Frame: Day 2
Population: Per Protocol Population: defined as all randomized subjects who satisfied the main inclusion / exclusion criteria, received investigational product, completed at least one treatment period, and did not present major violations to the protocol.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | LAS190792 5 µg (Part 1) | LAS190792 20 µg (Part 1) | LAS190792 50 µg (Part 1) | LAS190792 100 µg (Part 1) | LAS190792 200 µg (Part 1) | LAS190792 400 µg (Part 1) | Placebo (Part 1) | LAS190792 100 µg (Part 2) | LAS190792 400 µg (Part 2) | Tiotropium 18 μg | Indacaterol 150 μg | Placebo (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 36 | 35 | 37 | 37 | 37
Liters | -0.013 (0.333) | 0.161 (0.131) | 0.523 (0.448) | 0.536 (0.170) | 0.371 (0.333) | 0.599 (0.316) | 0.029 (0.144) | 1.369 (0.505) | 1.360 (0.472) | 1.379 (0.502) | 1.361 (0.481) | 1.338 (0.506)
Statistical Analysis 1: Comparison: LAS190792 100 µg (Part 2) vs Placebo (Part 2); Change from baseline to trough FEV1 was analyzed by means of an analysis of covariance (ANCOVA) for cross-over designs with sequence, treatment group and period as fixed effect factors, subject within sequence as random effect, and screening and baseline FEV1 value of each period as covariates; Test type: Superiority or Other; p < 0.0001, ANCOVA — All statistical comparisons were two-sided hypothesis tests, and the significance level was set at 0.05 without multiplicity adjustment; Least squares mean difference = 0.104, 95% CI 2-sided [0.060 to 0.149], Standard Error of Mean 0.023
Statistical Analysis 2: Comparison: LAS190792 400 µg (Part 2) vs Placebo (Part 2); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least squares mean difference = 0.178, 95% CI 2-sided [0.133 to 0.223], Standard Error of Mean 0.023

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Up to 36 hours after investigational product administration
Population: Pharmacokinetic population: defined as all randomized subjects who received at least one dose of investigational product in at least one treatment period and have evaluable PK parameters
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LAS190792 5 µg (Part 1) | LAS190792 20 µg (Part 1) | LAS190792 50 µg (Part 1) | LAS190792 100 µg (Part 1) | LAS190792 200 µg (Part 1) | LAS190792 400 µg (Part 1) | LAS190792 100 µg (Part 2) | LAS190792 400 µg (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 10
pg/mL | NA (NA) — With a lower limit of quantification (LLOQ) of 5 pg/mL, LAS190792 was not measurable in plasma following single doses of 5 µg | NA (NA) — With a LLOQ of 5 pg/mL, LAS190792 was not measurable in plasma following single doses of 20 μg, with the exception of one single sample (5.07 pg/mL) corresponding to a kinetic time-point of 0.5 h | 8.79 (4.86) | 19.5 (8.45) | 43.9 (16.8) | 59.7 (19.2) | 15.4 (6.39) | 56.2 (10.1)

4. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax)
Time Frame: Up to 36 hours after investigational product administration
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | LAS190792 5 µg (Part 1) | LAS190792 20 µg (Part 1) | LAS190792 50 µg (Part 1) | LAS190792 100 µg (Part 1) | LAS190792 200 µg (Part 1) | LAS190792 400 µg (Part 1) | LAS190792 100 µg (Part 2) | LAS190792 400 µg (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 10
Hours | NA [NA to NA] — With a lower limit of quantification (LLOQ) of 5 pg/mL, LAS190792 was not measurable in plasma following single doses of 5 µg | NA [NA to NA] — With a LLOQ of 5 pg/mL, LAS190792 was not measurable in plasma following single doses of 20 μg, with the exception of one single sample (5.07 pg/mL) corresponding to a kinetic time-point of 0.5 h. | 0.25 [0.25 to 0.5] | 0.5 [0.28 to 0.75] | 0.375 [0.25 to 0.5] | 0.517 [0.25 to 0.75] | 0.5 [0.25 to 0.75] | 0.517 [0.317 to 1.0]

5. Secondary Outcome: Area Under the Concentration-time Curve From Zero to the Time of the Last Measurable Concentration
Time Frame: Up to 36 hours after investigational product administration
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg.h/mL
Arm/Group | LAS190792 5 µg (Part 1) | LAS190792 20 µg (Part 1) | LAS190792 50 µg (Part 1) | LAS190792 100 µg (Part 1) | LAS190792 200 µg (Part 1) | LAS190792 400 µg (Part 1) | LAS190792 100 µg (Part 2) | LAS190792 400 µg (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 10
pg.h/mL | NA (NA) — With a lower limit of quantification (LLOQ) of 5 pg/mL, LAS190792 was not measurable in plasma following single doses of 5 µg | 0.106 (0.259) | 5.50 (3.53) | 20.1 (17.3) | 82.7 (43.3) | 122 (57.1) | 20.5 (15.4) | 127 (67.2)

ADVERSE EVENTS:
Time Frame: Up to 14 (±2) days after the last investigational product administration or after premature discontinuation.
Description: The Safety population comprised all randomised participants who received at least one dose of investigational product.
Arm/Group | LAS190792 5 µg (Part 1) | LAS190792 20 µg (Part 1) | LAS190792 50 µg (Part 1) | LAS190792 100 µg (Part 1) | LAS190792 200 µg (Part 1) | LAS190792 400 µg (Part 1) | Placebo (Part 1) | LAS190792 100 µg (Part 2) | LAS190792 400 µg (Part 2) | Tiotropium 18 μg | Indacaterol 150 μg | Placebo (Part 2)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/36 | 0/35 | 0/37 | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 2/6 | 3/6 | 1/6 | 2/6 | 2/6 | 4/6 | 3/12 | 4/36 | 9/35 | 6/37 | 15/37 | 11/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAS190792 5 µg (Part 1) (N=6) | LAS190792 20 µg (Part 1) (N=6) | LAS190792 50 µg (Part 1) (N=6) | LAS190792 100 µg (Part 1) (N=6) | LAS190792 200 µg (Part 1) (N=6) | LAS190792 400 µg (Part 1) (N=6) | Placebo (Part 1) (N=12) | LAS190792 100 µg (Part 2) (N=36) | LAS190792 400 µg (Part 2) (N=35) | Tiotropium 18 μg (N=37) | Indacaterol 150 μg (N=37) | Placebo (Part 2) (N=37)
Scrotal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAS190792 5 µg (Part 1) (N=6) | LAS190792 20 µg (Part 1) (N=6) | LAS190792 50 µg (Part 1) (N=6) | LAS190792 100 µg (Part 1) (N=6) | LAS190792 200 µg (Part 1) (N=6) | LAS190792 400 µg (Part 1) (N=6) | Placebo (Part 1) (N=12) | LAS190792 100 µg (Part 2) (N=36) | LAS190792 400 µg (Part 2) (N=35) | Tiotropium 18 μg (N=37) | Indacaterol 150 μg (N=37) | Placebo (Part 2) (N=37)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (3) | 3 (4) | 5 (7) | 6 (7) | 8 (8) | 4 (6)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 6 (6) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
In Part 1, many plasma concentrations at 50-100µg dose levels were BLOQ; thus only limited PK data were obtained for AUC(0-t), with plasma concentrations generally detected up to 1h post-administration; and at 200-400µg, up to 6 or 12h, respectively

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication and / or presentation whether complete or partial, of any part of the data or results of this study will not be allowed until global publication and study results disclosure by the sponsor as per EMA / FDA regulatory compliance obligations, and only after mutual agreement between the Investigator and AstraZemeca